CLINICAL TRIAL: NCT01136785
Title: Effects of Continuous Positive Airway Pressure (CPAP) Treatment on Glucose Control in Patients With Type 2 Diabetes
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0547
Record Dates: First submitted 2010-04-13; First posted 2010-06-03 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnea; Type 2 Diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active CPAP therapy (Active Comparator): 7 days of treatment in the laboratory with active CPAP therapy.
  Interventions: Device: active CPAP Therapy
- Sham CPAP therapy (Sham Comparator): 7 days of sham CPAP therapy in the laboratory.
  Interventions: Device: sham CPAP therapy

INTERVENTIONS:
Device: active CPAP Therapy — 7 days of active CPAP therapy
  Arms: Active CPAP therapy
Device: sham CPAP therapy — 7 days of sham CPAP therapy
  Arms: Sham CPAP therapy

SUMMARY:
The overall goal of the proposed protocol is to rigorously test the hypothesis that CPAP treatment has beneficial effects on glycemic control in patients with both type 2 diabetes (T2DM) and obstructive sleep apnea (OSA). If our hypothesis were to be proven, this would imply that CPAP treatment of OSA in patients with T2DM is an essential component of their glycemic control. The proposed work is thus expected to provide additional preventive and therapeutic approaches in the management of millions of patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with type 2 diabetes on a stable medication regimen (no change in diabetic medications in the previous 3 months) will be eligible.

Exclusion Criteria:

* Subjects on insulin will be excluded.
* Subjects with unstable cardiopulmonary disease, painful neuropathy, significant psychiatric illness, cognitive impairment and pregnancy will be excluded.
* Shift workers
* Subjects having traveled across >2 time zones less than one month prior to the study
* Diagnosis of a sleep disorder other than OSA by screening polysomnography
* Previous treatment with positive airway pressure or supplemental oxygen
* Requirement of supplemental oxygen or bi-level positive airway pressure for OSA treatment during titration
* Claustrophobia or other conditions of CPAP intolerance,
* Presence of active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago; Babak Mokhlesi, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Mokhlesi B, Grimaldi D, Beccuti G, Van Cauter E. Effect of one week of CPAP treatment of obstructive sleep apnoea on 24-hour profiles of glucose, insulin and counter-regulatory hormones in type 2 diabetes. Diabetes Obes Metab. 2017 Mar;19(3):452-456. doi: 10.1111/dom.12823. Epub 2016 Dec 12. PMID 27860160
- [Result] Mokhlesi B, Grimaldi D, Beccuti G, Abraham V, Whitmore H, Delebecque F, Van Cauter E. Effect of One Week of 8-Hour Nightly Continuous Positive Airway Pressure Treatment of Obstructive Sleep Apnea on Glycemic Control in Type 2 Diabetes: A Proof-of-Concept Study. Am J Respir Crit Care Med. 2016 Aug 15;194(4):516-9. doi: 10.1164/rccm.201602-0396LE. No abstract available. PMID 27525461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a 2:1 ratio (2 active CPAP: 1 sham CPAP), 22 eligible subjects who had completed baseline assessments underwent 1 week of in-laboratory active CPAP or sham CPAP therapy and completed the post-treatment assessments. Two subjects assigned to the CPAP group and one subject assigned to the sham group were excluded for protocol violations.
Groups:
- Active CPAP: 7 days of treatment in the laboratory with active CPAP.
  Continuous Positive Airway Pressure (CPAP) Therapy (active): CPAP is approved for the treatment of Obstructive Sleep Apnea
- Sham CPAP: 7 days of sham CPAP in the laboratory.
Period: Overall Study
Arm/Group | Active CPAP | Sham CPAP
Started | 15 | 7
Completed | 13 | 6
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Population: In a 2:1 ratio (2 active CPAP: 1 sham CPAP), 22 eligible subjects who had completed baseline assessments underwent 1 week of in-laboratory active CPAP or sham CPAP therapy and completed the post-treatment assessments. Two subjects assigned to the CPAP group and one subject assigned to the sham group were excluded for protocol violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CPAP | Sham CPAP | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.4) | 52.3 (3.1) | 55.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 4 | 2 | 6
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of 7-day Intervention in Mean Plasma Glucose Derived From 24 Hour Blood Sampling
Description: 24 hour blood sampling will be performed at baseline and at the end of the 7-day intervention. Glucose levels will be measured on each sample. Mean glucose level for all baseline samples will be calculated for each participant. Mean glucose levels for all samples collected at the end of the intervention will be calculated. Change in mean glucose level from baseline to end of intervention will be calculated for each participant.
Time Frame: after 1 week of CPAP therapy in the laboratory
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 13 | 6
mg/dl | -13.7 (3.6) | -2.9 (1.4)
Statistical Analysis 1: Comparison: Active CPAP vs Sham CPAP; two-sided t test for the change from baseline between the treated and untreated groups; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

2. Primary Outcome: Change From Baseline in Mean Glucose From Continuous Interstitial Glucose Monitoring Over 36-40 Hours
Description: Continuous Glucose monitoring will provide interstitial glucose levels for 36-40 hours at baseline and after one week of active or sham CPAP therapy. The mean glucose level of all samples collected at baseline will be calculated for each participant. The mean glucose level of all samples collected at the end of the 7-day intervention will be calculated for each participant. For each participant, we will calculate the change in mean glucose level from baseline till end of the intervention.
Time Frame: change in mean interstitial glucose after 1 week of active or sham CPAP therapy in the laboratory
Population: Due to sensor failures, valid profiles of interstitial glucose were available in 10 participants with the active CPAP group and 4 participants in the sham CPAP group.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 10 | 4
mg/dL | -12.4 (3.9) | 1.5 (2.2)
Statistical Analysis 1: Comparison: Sham CPAP; comparing pre and post Interstitial Glucose levels in the active CPAP group; Test type: Superiority or Other; p = 0.011, 2-sided Paired t-test

3. Primary Outcome: Change in Mean Serum Insulin Derived From 24 Hour Blood Sampling
Description: Serum insulin levels will be measured on each sample collected during 24-h sampling at baseline and at the end of the 7-day intervention. Mean insulin level over 24 hours will be calculated for each participant at baseline and at the end of the intervention. For each participant, we will calculate the change in mean insulin level from baseline.
Time Frame: after 1 week of therapy in the laboratory
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- CPAP: 7 days of sham CPAP in the laboratory.
Arm/Group | Active CPAP | CPAP
Number analyzed (Participants) | 13 | 6
pmol/L | -25.8 (16.5) | 28.4 (21.6)
Statistical Analysis 1: Comparison: Active CPAP vs CPAP; Test type: Superiority or Other; p = 0.071, t-test, 2 sided

4. Secondary Outcome: Change in Mean Plasma Cortisol Level From 24-h Sampling
Description: The mean plasma cortisol level will be calculated for all samples collected at baseline and for all samples collected at the end of the intervention in participants randomized to the active CPAP arm. The goal of the analysis of cortisol, growth hormone and norepinephrine levels was to explore putative mechanisms underlying the effects of active CPAP therapy. Examining putative hormonal mechanisms underlying changes in glucose levels in the sham CPAP arm was not part of our aims. For each participant, the change in mean cortisol level from baseline to end of intervention will be calculated.
Time Frame: after 1 week of active CPAP therapy in the laboratory
Measure: Mean (95% Confidence Interval); unit: microgram/dL
Groups:
- Active CPAP: The goal of the present analysis is to explore mechanisms by which CPAP therapy led to improvement in the 24-h glucose levels. We focus on the 12 participants who had complete 24-h profiles of glucose, insulin and counter-regulatory hormones before and after treatment with active CPAP.
Arm/Group | Active CPAP
Number analyzed (Participants) | 12
microgram/dL | -0.1 [-0.8 to 0.7]
Statistical Analysis 1: Comparison: Active CPAP; Plasma cortisol pre and post 1-week of active CPAP; Test type: Superiority or Other; p = 0.754, two-sided paired t-test

5. Secondary Outcome: 24-hr Profile of Plasma Growth Hormone
Description: The mean plasma growth hormone level will be calculated for all samples collected at baseline and for all samples collected at the end of the intervention in participants randomized to the active CPAP arm. The goal of the analysis of cortisol, growth hormone and norepinephrine levels was to explore putative mechanisms underlying the effects of active CPAP therapy. Examining putative hormonal mechanisms underlying changes in glucose levels in the sham CPAP arm was not part of our aims. For each participant, the change in mean cortisol level from baseline to end of intervention will be calculated.
Time Frame: after 1 week of active CPAP therapy in the laboratory
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Active CPAP
Number analyzed (Participants) | 12
ng/ml | -0.02 [-0.15 to 0.04]
Statistical Analysis 1: Comparison: Active CPAP; comparing pre and post levels in the active CPAP group; Test type: Superiority or Other; p = 0.308, two-sided paired t-test

6. Secondary Outcome: Change in 24-h Mean Level of Plasma Norepinephrine
Description: The mean plasma norepinephrine level will be calculated for all samples collected at baseline and for all samples collected at the end of the intervention in participants randomized to the active CPAP arm. The goal of the analysis of cortisol, growth hormone and norepinephrine levels was to explore putative mechanisms underlying the effects of active CPAP therapy. Examining putative hormonal mechanisms underlying changes in glucose levels in the sham CPAP arm was not part of our aims. For each participant, the change in mean norepinephine level from baseline to end of intervention will be calculated.
Time Frame: after 1 week of active CPAP therapy in the laboratory
Measure: Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Active CPAP: The goal of the present analysis is to explore mechanisms by which CPAP therapy led to improvement in the 24-h glucose levels. We focus on the 8 participants who had complete 24-h profiles of plasma norepinephrine before and after treatment with active CPAP.
Arm/Group | Active CPAP
Number analyzed (Participants) | 8
pg/ml | -60.9 [-124.7 to -6.2]
Statistical Analysis 1: Comparison: Active CPAP; comparing pre and post levels in the active CPAP group; Test type: Superiority or Other; p = 0.036, two-sided paired t-test

ADVERSE EVENTS:
Arm/Group | Active CPAP | Sham CPAP
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 0/7

LIMITATIONS AND CAVEATS:
One limitation of the study is that two subjects assigned to sham CPAP received defective sham devices that delivered therapeutic pressure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes